CLINICAL TRIAL: NCT07087093
Title: Effects of Ketone Esters on Circulating Senescent T Lymphocytes (T Cells) and Inflammation Levels in the Elderly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ketone Esters-2024214
Record Dates: First submitted 2025-03-24; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: The Elderly
Keywords: ketone ester; the eldly; Senescent T cell; inflammatory factors
MeSH Terms: interventions — formic acid 4-(3-oxobutyl)phenyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ketone ester group (Experimental)
  Interventions: Other: Ketone ester

INTERVENTIONS:
Other: Ketone ester — KetoneAid Ke4 Pro Ketone Ester：20ml, tid po

SUMMARY:
Studies have shown that aging can promote a variety of pathological processes, such as myocardial remodeling and cardiac dysfunction caused by ischemia-reperfusion injury and pressure load. Previous studies found that the level of circulating beta-hydroxybutyric acid decreased significantly with age. It has been reported that the ketogenic diet reduces the occurrence of tumors and neurodegenerative diseases in mice, improves motor coordination and endurance, and ultimately extends life span. Current research results have confirmed that ketone bodies have multiple mechanisms to exert beneficial effects on cardiovascular diseases. However, the effect of age-related cardiovascular disease has not been reported.

In order to further clarify the role of beta-hydroxybutyric acid in age-related cardiovascular diseases, find new intervention targets for elderly cardiovascular diseases, and develop new effective prevention and treatment measures for elderly cardiovascular diseases. We will further investigate this hypothesis by establishing a clinical cohort of the elderly population.

DETAILED DESCRIPTION:
It is predicted that by 2050, the total number of people over 65 years old in China will reach 400 million (accounting for 26.9% of the total population), and the number of people over 80 years old will reach 150 million. Population aging is the main driving force of cardiovascular diseases, and cardiovascular diseases in the elderly will become a major clinical problem threatening the health of our people and a social problem involving people's livelihood. Therefore, it is an important research direction in the cardiovascular field to deeply explore the pathogenesis of elderly cardiovascular diseases and find effective prevention and control targets.

Studies have shown that aging can promote a variety of pathological processes, such as myocardial remodeling and cardiac dysfunction caused by ischemia-reperfusion injury and pressure load. Previous studies found that the level of circulating beta-hydroxybutyric acid decreased significantly with age. It has been reported that the ketogenic diet reduces the occurrence of tumors and neurodegenerative diseases in mice, improves motor coordination and endurance, and ultimately extends life span. Current research results have confirmed that ketone bodies have multiple mechanisms to exert beneficial effects on cardiovascular diseases. However, the effect of age-related cardiovascular disease has not been reported.

In order to further clarify the role of beta-hydroxybutyric acid in age-related cardiovascular diseases, find new intervention targets for elderly cardiovascular diseases, and develop new effective prevention and treatment measures for elderly cardiovascular diseases. We will further investigate this hypothesis by establishing a clinical cohort of the elderly population.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 65~80 years old.
2. The subjects are in good health, and no history of chronic diseases.

Exclusion Criteria:

1. Have used immunosuppressants or hormone drugs in the past six months.
2. There has been a significant change in diet within the past month.
3. Having digestive tract surgery within one year.
4. Severe liver dysfunction (alanine aminotransferase level > 3.0 upper limit of normal).
5. Severe kidney dysfunction (creatinine clearance rate < 30 mL/min).
6. History of malignant tumor.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
T cell senescence level (Protein 53、Protein 21 and Protein 16) | From enrollment to the end of treatment at 2 weeks
  Expression of protein 53、protein 21 and protein 16 in human plasma used by western blot.

SECONDARY OUTCOMES:
Circulating inflammatory factor levels (monocyte chemoattractant protein-1 and interleukin-6) | From enrollment to the end of treatment at 2 weeks
  Expression of monocyte chemoattractant protein-1 and interleukin-6 in human plasma used by enzyme linked immunosorbent assay.
Ankle-brachial index | From enrollment to the end of treatment at 2 weeks
  The ankle-brachial index value was measured by dopplex ankle-brachial index detector.

OTHER OUTCOMES:
Ejection fraction (EF) levels | From enrollment to the end of treatment at 2 weeks
  Use cardiac echocardiography to assess the ejection fraction level
NT-proBNP level | From enrollment to the end of treatment at 2 weeks
  NT-proBNP level was used by chemiluminescence immunoassay.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No